CLINICAL TRIAL: NCT05911347
Title: Effect of Modified Cellulose on Colonic Fermentation of Inulin (COCOA2)
Brief Title: Effect of Modified Cellulose on Colonic Fermentation of Inulin
Acronym: COCOA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FMHS 19-0622
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAP; Inulin; Psyllium; Cellulose
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psyllium; Methylcellulose; maltodextrin

STUDY DESIGN:
Intervention Model Description: 3 way cross-over
Who Masked: Participant, Outcomes Assessor
Masking Description: Test meals will have similar appearance and flavour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psyllium (Active Comparator): Psyllium 15 g+ inulin 15 gm in 375ml water
  Interventions: Dietary Supplement: Psyllium
- maltodextrin (Placebo Comparator): Maltodextrin 15 g + inulin 15 gm in 375 ml water
  Interventions: Dietary Supplement: Maltodextrin
- Methylcellulose (Experimental): Methylcellulose 15g + Inulin 15 g in 375 ml water
  Interventions: Dietary Supplement: Methylcellulose

INTERVENTIONS:
Dietary Supplement: Psyllium — 15g psyllium added to inulin solution to form a gel
  Arms: Psyllium
Dietary Supplement: Methylcellulose — 15 g methylcellulose added to inulin solution to form a gel
  Arms: Methylcellulose
Dietary Supplement: Maltodextrin — 15g maltodextrin added to inulin solution to form a gel
  Arms: maltodextrin

SUMMARY:
A 3-way randomised cross-over study to test the hypothesis that combining either psyllium or methylcellulose to form a gel incorporating inulin will reduce gas production as compared to inulin given with a placebo, maltodextrin. Subjects will attend on 3 separate days separated by a minimum of one week an consume one of 3 test meals. Serial breath samples with be obtained to measure hydrogen and methane over the next 24 hours. Primary endpoint: Area under curve (AUC) from time 0-6 hours (AUC 0-6) of breath hydrogen (ppm.hour) after treatment intake. The investigators will also assess whole gut transit time using the blue muffin and correlate breath hydrogen production with in vitro fermentation results.

DETAILED DESCRIPTION:
A 3-way randomised cross-over study to test the hypothesis that combining either psyllium or methylcellulose to form a gel incorporating inulin will reduce gas production as compared to inulin given with a placebo, maltodextrin. Subjects will attend on 3 separate days separated by a minimum of one week an consume one of 3 test meals. Serial breath samples with be obtained to measure hydrogen and methane over the next 24 hours.

Primary endpoint: Area under curve (AUC) from time 0-6 hours (AUC 0-6) of breath hydrogen (ppm.hour) after treatment intake. Whole gut transit time will be assessed from the time that stool turns blue after ingestion of a muffin labelled with blue food colouring.

Secondary endpoint:

1. AUC (0-24h) breath hydrogen / methane
2. Oro-cecal transit time and whole gut transit time.
3. Gas production/ metabolites/ microbiota during in vitro fermentation studies at Quadram
4. Effect of habitual dietary FODMAPs intake on breath hydrogen response to inulin.

The interventions will be dietary interventions, using all food grade materials (sugars and fibres) provided in commonly used doses:

Breath hydrogen will be correlated with in vitro carbohydrate fermentation profile assessed using stool samples collected before intervention

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older.
* Able to give informed consent.
* Scoring ≤5 (i.e., mild, or less) for symptoms of flatulence, bloating, abdominal pain, loose stool, and hard stool in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
* Agrees to consume the meals provided.
* Agrees to not smoke during the breath sampling period.

Exclusion Criteria:

* Pregnancy declared by candidate.
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
* Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
* Intestinal stoma.
* Any medical condition making participation potentially compromising participation in the study e.g., diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
* Will not agree to dietary restrictions required.
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
* Participants who are taking antibiotics or probiotics as it might alters gut microbiota.
* Poor understanding of English language.
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Breath hydrogen | 0-6 hoursafter ingestion
  AUC 0-6 hours after ingestion

SECONDARY OUTCOMES:
Breath hydrogen | 0-24 hours post ingestion
  AUC 0-24 hours
Breath methane | 0-24 hours post ingestion
  AUC 0-24 hours
Transit time | Whole gut transit measured once before intervention
  whole gut transit time

CONTACTS AND LOCATIONS:
Overall Officials: Robin D Spiller, MD, Principal Investigator — University of Nottingham
Locations (1):
- University Hospital Clinical Research Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunn D, Abbas Z, Harris HC, Major G, Hoad C, Gowland P, Marciani L, Gill SK, Warren FJ, Rossi M, Remes-Troche JM, Whelan K, Spiller RC. Psyllium reduces inulin-induced colonic gas production in IBS: MRI and in vitro fermentation studies. Gut. 2022 May;71(5):919-927. doi: 10.1136/gutjnl-2021-324784. Epub 2021 Aug 5. PMID 34353864
- [Derived] Reid JESJ, Alhasani AT, MacCalman T, Amor D, Aliyu AI, Modasia AA, Harris H, Warren FJ, Hoad C, Gowland PA, Yakubov GE, Crooks C, Corsetti M, Marciani L, Spiller RC. A randomised, placebo-controlled trial in healthy humans of modified cellulose or psyllium evaluating the role of gelation in altering colonic gas production during inulin co-administration. Food Funct. 2026 Feb 4. doi: 10.1039/d5fo03532e. Online ahead of print. PMID 41636227